CLINICAL TRIAL: NCT06430177
Title: The Effect of Sujok Therapy on Patient Comfort, Pain Intensity, and Anxiety Level in Cancer Patients With Port Catheter Placement: A Randomized, Placebo and Controlled Study
Brief Title: The Effect of Sujok Therapy on Patient Comfort, Pain Intensity, and Anxiety Level in Cancer Patients With Port Catheter Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/07-28
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Chemotherapy Effect
Keywords: Su Jok; Pain; Anxiety
MeSH Terms: conditions — Neoplasms; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Su Jok will be done
  Interventions: Behavioral: Su Jok
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Su Jok — Su Jok will be done
  Arms: Experimental

SUMMARY:
Cancer is a fatal disease characterized by uncontrolled growth and proliferation of tissues and organs in the human body. Among cancer treatments, chemotherapy is the most commonly used treatment method. The drugs used in chemotherapy cause vascular toxic effects during administration, frequent blood samples taken from the patient, antibiotic treatments applied, parenteral nutrition treatments. Subcutaneous venous port catheter (SCVPK), which is a permanent and long-term vascular access route that can be used for medical purposes and in emergency situations, is a frequently preferred and safe intravenous access route because it is not visible outside the body, is well tolerated by the patient, and has a low risk of infection. However, invasive procedures such as port needle insertion and replacement can also cause pain, anxiety and changes in vital signs in patients. Nowadays, the use of non-pharmacological approaches as well as pharmacological methods is increasing in the management of symptoms such as anxiety before the invasive procedure and pain during application in patients receiving chemotherapy treatment. These approaches improve the quality of life of patients and have a positive physiological effect. One of these approaches is sujok therapy. In Su Jok application; The reflection points of the organs are on the hands and feet. These points reflect to the body organ in that area and healing occurs. By finding the right point, energy flow is provided by massaging with appropriate applicators. This research will be conducted to examine the effect of Sujok therapy on pain intensity and anxiety level in cancer patients who have undergone port catheter placement.

The research will be conducted as a randomized experimental and placebo study with a pretest-posttest control group in the oncology service of Fethi Sekin City Hospital. 90 (30 experimental, 30 control, 30 placebo) cancer patients who accept the research and meet the sample criteria of the study will be subjected to port catheter application. Application areas for pain, anxiety and stress before the port catheter to the patients in the experimental group will be determined with the help of a probe (diagnostic stick), and seeds will be added to these points approximately 45 minutes before the application and fixed with a patch. For cancer patients in the placebo group, the same procedure will be performed with seeds that have a neutral effect on the body. No procedure will be applied to the patients in the control group. Patient Information Form, General Comfort Scale (GAS), Visual Analog Scale -Pain (VAS-P), Visual Analog Scale -Anxiety (VAS-A) and State-Trait Anxiety Scale were used as data collection tools. (DSKÖ) scale will be used. SPPS 21.0 (Statistical Programme for Social Sciences) package program will be used to evaluate the data obtained from the research. It is thought that if the objectives of the study are achieved, it will help reduce the level of pain and anxiety that may occur during and after port catheter application. In addition, it will contribute to the professional advancement of the project manager, which is a career development project. The positive results in this study will guide other interventions to increase the comfort level of cancer patients who will undergo port catheterization and reduce the level of pain and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Ability to communicate adequately
* Being diagnosed with cancer
* Will receive chemotherapy treatment
* Port catheter placement will be performed
* Suitable for Implantable Port Catheter Placement

Exclusion Criteria:

* Loss of sensation in the hands, amputation, injury, etc. that would prevent practice. to be
* Patients with chronic pain or anxiety disorders, using any analgesics or anxiolytics

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
General Comfort Scale | two hours later
  It is a four-point Likert type consisting of 48 items to measure the expected comfort result of the patient in order to test the taxonomic structure created after completing the conceptual studies of comfort. In this research, the scale adapted to Turkish by Kuğuoğlu and Karabacak was used. The scale is a four/six point Likert type and contains a total of 48 items. A four-point Likert type was preferred in the study due to its ease of use. Scale sub-dimensions; relief (16 items), relaxation (17 items) and overcoming problems (15 items). The response patterns of the scale, which consists of positive and negative items, are given in mixed order. Accordingly, in positive statements, a high score (4p) indicates high comfort, a low score (1p) indicates low comfort, in negative items, a low score (1p) indicates high comfort, and a high score (4p) indicates low comfort. In the evaluation of the scale; The negative scores obtained are reverse coded and added to the positive items.
Visual Analog Scale - Anxiety | two hours later
  The patients were asked to measure their anxiety level during rest or activity on a 10 cm long horizontal line.
  is requested to show. The value 0 is at the beginning of the line and 10 is at the end. 10 indicates extreme anxiety, 0 indicates not at all.
  It shows that there is no concern. VAS scale is used quite frequently during the evaluation of anxiety severity.
  is used
Visual Analog Scale -Agrı | two hours later
  It is used to convert some values that cannot be measured numerically into numerical values. Two extreme definitions of the parameter to be evaluated are written at both ends of a 100 mm line, and the patient is asked to indicate where his/her situation is appropriate on this line by drawing a line, placing a dot, or pointing.
State-Trait Anxiety Scale | two hours later
  It is a scale developed to measure individuals' state and trait anxiety levels. It is a self-assessment scale whose Turkish validity and reliability studies have been conducted. In this study, the section of the scale measuring state anxiety was used to determine the state anxiety levels of the patients. State Anxiety Scale is a 4-point Likert type with 20 items and is scored according to the severity of the feelings, thoughts or behaviors expressed by the items as "not at all": 1, "somewhat": 2, "a lot": 3, "completely": 4. . The scale includes directly or reverse scored expressions.

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat university, Elâzığ, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after it is finished